CLINICAL TRIAL: NCT06688097
Title: Ultrasound-Guided Esophageal Compression During Adult Mask Ventilation: A Prospective Observational Study
Brief Title: Ultrasound-Guided Esophageal Compression During Adult Mask Ventilation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Han (Other)
Responsible Party: Sponsor-Investigator, Liu Han, Director, Department of Anesthesia, Pain and Perioperative Medicine, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KY20240924-01
Record Dates: First submitted 2024-10-15; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Laparoscopic Surgery; Ultrasonography; Compression of Esophagus; Stomach Distended
MeSH Terms: conditions — Gastric Dilatation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Control Group) (No Intervention): No esophageal compression is applied, and FMV is performed for 4 minutes.
- Group B (Intervention Group) (Experimental): Ultrasound-guided esophageal compression plus FMV: before the start of FMV, ultrasound is used to locate the esophagus, and pressure is applied to the esophagus at the cricoid level to collapse the esophageal lumen. Esophageal pressure is released just before tracheal intubation following 4 minutes of ventilation.
  Interventions: Behavioral: Compression of esophageal

INTERVENTIONS:
Behavioral: Compression of esophageal — Before the start of FMV, ultrasound is used to locate the esophagus, and pressure is applied to the esophagus at the cricoid level to collapse the esophageal lumen. Esophageal pressure is released just before tracheal intubation following 4 minutes of ventilation.
  Arms: Group B (Intervention Group)

SUMMARY:
A total of 103 elective surgery patients who met the inclusion criteria were selected. After screening for eligibility according to the inclusion and exclusion criteria and signing informed consent, they were randomly divided into two groups. Upon entering the operating room, routine ECG monitoring was initiated, and a peripheral vein was opened. Ultrasound was used to measure the baseline cross-sectional area (CSA) of the gastric antrum in the supine position. After general anesthesia induction, positive pressure ventilation was applied via face mask. Group A received no external compression, while Group B underwent esophageal compression under ultrasound guidance.

DETAILED DESCRIPTION:
Upon entering the operating room, intravenous access is established, and oxygen is administered. Standard vital sign monitoring is initiated, including heart rate, non-invasive blood pressure, peripheral oxygen saturation, temperature monitoring, and BIS monitoring. Ultrasound is used to measure the cross-sectional area (CSA) of the gastric antrum before the onset of FMV.

Oxygen is administered via face mask for denitrogenation, with 100% pure oxygen (6 L/min flow rate). Intravenous medications are sequentially administered: midazolam 0.03 mg/kg, propofol 1-2 mg/kg, sufentanil 0.5 μg/kg, remifentanil 1 μg/kg, and rocuronium bromide 0.6 mg/kg. After the patient loses consciousness and the eyelash reflex is absent, FMV is initiated. The trial employs a pressure-controlled ventilation (PCV) mode with a pressure of 18 cmH2O, a level sufficient to provide adequate alveolar ventilation while staying below the threshold for significant gastroesophageal regurgitation. The respiratory rate is set at 14 breaths per minute with an inspiration-to-expiration ratio of 1:2.

After three minutes of FMV, the gastric antrum CSA is measured again in supine, semi-recumbent, and right lateral decubitus positions. Video laryngoscopy is used to record POGO scores before and after ultrasound-guided esophageal compression, and after 4 minutes of ventilation, tracheal intubation is performed. Grouping:

Group A (Control Group): No esophageal compression is applied, and FMV is performed for 4 minutes.

Group B (Intervention Group): Ultrasound-guided esophageal compression plus FMV: before the start of FMV, ultrasound is used to locate the esophagus, and pressure is applied to the esophagus at the cricoid level to collapse the esophageal lumen. Esophageal pressure is released just before tracheal intubation following 4 minutes of ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* American Society of Anesthesiologists (ASA) Physical Status Classification I-II.
* Body Mass Index (BMI) between 18 and 28 kg/m².
* Patients undergoing elective tracheal intubation for general anesthesia.
* Patients scheduled for laparoscopic surgery.
* Fasting for ≥8 hours and abstaining from liquids for ≥2 hours before surgery, with low risk of gastroesophageal regurgitation and aspiration.

Exclusion Criteria:

* Suspected difficult FMV (e.g., age >55 years, BMI >26 kg/m², edentulous, history of snoring, and long beard; presence of two or more factors).
* Pre-existing respiratory, pharyngeal, laryngeal, facial, or neck pathology.
* History of gastrointestinal surgery, gastroesophageal reflux disease (GERD), or high risk of aspiration.
* Severe cardiac, cerebral, pulmonary, hepatic, or renal diseases.
* Patients requiring non-invasive ventilation prior to surgery.
* Patients currently participating in other clinical trials or who refuse to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of gastric distension | During anesthesia induction
  Defined as a significant increase in gastric antrum CSA with acoustic shadowing or the characteristic "comet-tail sign," or when the enlarged gastric antrum obstructs the surgical field

SECONDARY OUTCOMES:
The positional relationship between the esophagus and trachea | Before anesthesia induction
  Observe the position of the esophagus relative to the trachea without the application of pressure on the patient, and assess whether there is any positional change of the esophagus relative to the trachea under ultrasound guidance after esophageal compression, ensuring the accuracy and safety of esophageal compression.
Tidal volume | During anesthesia induction
  Observe whether tidal volume is affected after ultrasound-guided esophageal compression and evaluate the impact of esophageal compression on ventilation quality. Effective esophageal compression should maintain a tidal volume of no less than 6 ml/kg for the patient.
Oxygen saturation | During anesthesia induction
  Observe whether oxygen saturation is affected after ultrasound-guided esophageal compression and evaluate the impact of esophageal compression on ventilation quality. Effective esophageal compression should maintain the patient's oxygen saturation at no less than 95%.
Airway plateau | During anesthesia induction
  Observe the values of airway plateau pressure during esophageal compression to evaluate the mechanical impact of esophageal compression on the airway. An airway plateau pressure not exceeding 20-25 cmH₂O indicates effective esophageal compression.
The percentage of glottic opening (POGO) score | During tracheal intubation, immediately
  The percentage of glottic opening (POGO) score represents the portion of the glottis visualized. It is defined anteriorly by the anterior commissure and posteriorly by the interarytenoid notch. The score ranges from 0% when none of the glottis is seen to 100% when the entire glottis including the anterior commissure is seen.
  A POGO score of 100% denotes visualization of the entire glottic opening in linear fashion from the anterior commissure to the posterior cartilages . If none of the glottic opening is seen, then the POGO score is 0%. The higher the POGO value, the less impact effective esophageal compression has on ventilation performance.
Surgeon's evaluation of gastric insufflation | Upon the start of surgery, immediately
  The degree of gastric distention is assessed by the same surgeon through laparoscopy. A score of 0 is given when there is no significant gastric distention, a score of 1 is given when there is noticeable gastric distention that does not affect the surgical procedure, and a score of 2 is given when there is significant gastric distention that affects the surgery, requiring the placement of a gastric tube for decompression. The number of postoperative vomiting episodes is recorded: 0 episodes is scored as 0, 1-2 episodes is scored as 1, and more than 2 episodes is scored as 2. A lower score indicates better esophageal compression effectiveness.
Rate of esophageal diameter change | During anesthesia induction
  Compare the diameter before and after esophageal compression and calculate the percentage change in diameter. After esophageal compression, the diameter of the esophagus should decrease. The percentage change in diameter is usually expressed as a negative value, indicating that the esophagus has constricted after compression. If the percentage change is positive, it suggests that the compression effect is not ideal, and the esophagus may not have been effectively compressed.
Esophageal compression pressure | During anesthesia induction
  Recording esophageal compression pressure can ensure that the applied pressure is within an effective range, help understand the relationship between compression intensity and ventilation efficacy, and promptly identify potential complications, such as airway compression or esophageal injury caused by excessive pressure, allowing for necessary interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No